CLINICAL TRIAL: NCT01923545
Title: Multi-Center, Randomized, Open, Phase II Study to Evaluate Efficacy and Safety in Chemotherapy-induced Neutropenia of Once-per-cycle DA-3031(PEG-G-CSF) and Daily G-CSF in Patients With Malignancies Receiving Myelosuppressive Chemotherapy
Brief Title: Phase II Study of DA-3031(PEG-G-CSF) in Chemotherapy-induced Neutropenia
Acronym: PEG-G-CSF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA3031_NP_II
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Chemotherapy Induced Neutropenia
Keywords: PEG-G-CSF
MeSH Terms: interventions — pegylated granulocyte colony-stimulating factor, human; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- DA-3031 3.6mg (Experimental): PEG-G-CSF
  Interventions: Drug: PEG-G-CSF
- DA-3031 6mg (Experimental): PEG-G-CSF
  Interventions: Drug: PEG-G-CSF
- Leucostim® (Active Comparator): G-CSF
  Interventions: Drug: G-CSF

INTERVENTIONS:
Drug: PEG-G-CSF — Vial, 3.6mg/day or 6mg/day, single dosing per cycle, for 1 cycle
  Other Names: DA-3031
  Arms: DA-3031 3.6mg; DA-3031 6mg
Drug: G-CSF — Vial, 100ug/m2/day, multiple dosing per cycle(daily administration, up to 10 days), for 1 cycle
  Other Names: Leucostim®
  Arms: Leucostim®

SUMMARY:
This study is to examine which dose of DA-3031(PEG-G-CSF) has similar efficacy and safety compared to daily G-CSF in chemotherapy-induced neutropenia.

DETAILED DESCRIPTION:
Eligible subjects are randomly assigned to receive once-per-cycle DA-3031(PEG-G-CSF) or daily G-CSF(up to 10 days). This study is conducted for 1 cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of stage II or III breast cancer
2. Age : ≥18, ≤70
3. TAC regimen as adjuvant therapy
4. ANC≥1,500/mm3, Platelet≥100,000/mm3, ECOG : 0 or 1
5. Creatinine < 1.5 x ULN
6. Total bilirubin/AST/ALT < 1.5 x ULN, ALP < 2.5 x ULN
7. Have given a written, informed consent

Exclusion Criteria:

1. Received any other investigational drugs within 30 days of informed consent date
2. Received systemic antibiotics within 72 hours of chemotherapy into this study or Radiation therapy within 4 weeks of informed consent date
3. Infective symptom before chemotherapy into this study
4. Pregnant or lactating women
5. Prior bone marrow or stem cell transplantation
6. Other malignancy history within 5 years
7. HIV positive
8. Prior exposure to pegfilgrastim or filgrastim or other colony-stimulating factors within 6 weeks of informed consent date
9. Prior chemotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Duration of grade 4 neutropenia in cycle 1 | 21 day
  Grade 4 neutropenia means the ANC count is less than 500/mm3.

SECONDARY OUTCOMES:
ANC nadir in cycle 1 | 21 day
  ANC nadir means the lowest point of ANC count.
Time to ANC recovery in cycle 1 | 21 day
  ANC recovery means the ANC count is more than 2,000/mm3.
Incidence of febrile neutropenia in cycle 1 | 21 day
  Febrile neutropenia means the ANC count is less than 1,000/mm3 and body temperature is more than 38.5 degrees celsius.
Incidence of IV antibiotics administration in cycle 1 | 21 day
  IV antibiotics administration means that antibiotics are administered through intravenous route.

CONTACTS AND LOCATIONS:
Overall Officials: JaeHong Seo, M.D., Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University GURO hospital, Seoul, South Korea